CLINICAL TRIAL: NCT00709514
Title: A Phase II, Double-blind, Placebo-controlled Clinical Evaluation of DCB-WH1 in Healing of Chronic Diabetic Foot Ulcers
Brief Title: Clinical Evaluation of DCB-WH1 in Healing of Chronic Diabetic Foot Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCB-WH1-CP001
Record Dates: First submitted 2008-06-27; First posted 2008-07-03 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Diabetic Foot Ulcer
Keywords: Oneness; DCB-WH1; DCB-WH1-CP001; chronic; diabetic; foot ulcers; topical ointment
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Foot Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DCB-WH1 ointment (Experimental): DCB-WH1 ointment 1.25%, topical use, two times daily for 12 weeks or until ulcer closes completely or discontinuation due to treatment failure, whichever comes first.
  Interventions: Drug: DCB-WH1 ointment
- Placebo (Placebo Comparator): Placebo, topical use, two times daily for 12 weeks or until ulcer closes completely or discontinuation due to treatment failure, whichever comes first.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DCB-WH1 ointment — DCB-WH1 ointment (1.25%), topically applied twice daily
  Arms: DCB-WH1 ointment
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this Phase 2 study is to evaluate the efficacy of DCB-WH1 ointment in wound closure as compared to vehicle control when applied topically to chronic diabetic foot ulcers for 12 weeks. The secondary objective of this study is to collect safety information of DCB-WH1 ointment.

This is a randomized, double-blind, parallel group, vehicle-controlled, multi-center study of DCB-WH1 ointment applied topically to grade 1 foot ulcers (according to Wagner grading system) in 50 subjects with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 20 or older with diabetes mellitus (Type 1 or 2) who has a cutaneous ulcer on the foot and present for at least 2 weeks
2. The target ulcer is classified as a grade 1 ulcer according to a modified Wagner system, which includes wounds involving the epidermis, the dermis, the hypodermis or the subcutaneous fat but not the tendon or joint capsule. The thickness of aforesaid layers wounds be approximately between 0.2 mm and 8 mm and is ranging in size between 3 and 15 cm2 post debridement.
3. An ankle brachial index ≥0.80.
4. The study ulcer should show "infection control" as judged by the investigator
5. The subject should be free of any necrotic or infected soft and bony tissue.
6. Signed informed consent form.

Exclusion Criteria:

1. Ulcers caused by venous or arterial insufficiency, osteomyelitis.
2. Poor nutritional status (albumin < 3g/dl), poor diabetic control (HbA1c > 10%), anemia (hemoglobin<10 g/dL), a leukocyte counts < 1,000/cumm.
3. Requiring prostaglandin treatment.
4. Requiring treatment with corticosteroids, immunosuppressive or chemotherapeutic agents, radiotherapy.
5. Presence of necrosis, purulence or sinus tracts that cannot be removed by debridement.
6. Presence of connective tissue disease, renal failure (*eGFR≦30 ml/min/1.73m2), abnormal liver function (Aspartate Aminotransferase(AST), Alanine Aminotransferase(ALT)>2.5x upper limit of normal range), malignancy.
7. vascularization surgery performed <8 weeks before entry in the study.
8. A history of cerebrovascular events, coronary intervention (stent or coronary artery bypass graft (CABG)) or myocardial infarction, within 6 months prior to study.
9. Female patient who has a positive pregnancy test or who is breastfeeding or unwilling to use appropriate contraceptive methods during study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-12; Primary Completion 2011-04 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The incidence of complete ulcer closure | 12 weeks

SECONDARY OUTCOMES:
The time of healing rate and change in ulcer area | 12 weeks
  time to ulcer closure, time to half ulcer closure, ulcer closure rate at endpoint, change and percentage change from baseline in ulcer size

CONTACTS AND LOCATIONS:
Overall Officials: Low-Tong Ho, MD, Principal Investigator — Taipei Veterans General Hospital Taipei
Locations (1):
- Clinical Research Division, Taipei, Taiwan